CLINICAL TRIAL: NCT00759382
Title: Prognostic Role of Primary Non Small Cell Lung Carcinoma Standardized F18-FDG Uptake Values (SUV and TLG) Measured With F18-fluorodeoxyglucose Positron Emission Tomography (F18-FDG-PET): a Non Interventional Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Other Study IDs: 01071
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non small cell lung carcinoma; PET scan; Observational study; Non metastatic; treated; curative intent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Patients with non-small cell lung carcinoma treated with curative intent

SUMMARY:
The primary aim of this non interventional study is to assess the independent prognostic role on overall survival of primary tumour 18F-FDG uptake value (SUVmax) measured on 18fluorodeoxyglucose positron emission tomography (18F-FDG-PET) in patients with non-metastatic non-small cell lung cancers treated with curative intent, taking into account the other conventional prognostic factors (performance status, age, sex, disease stage).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically demonstrated NSCLC
* Stage I-III treated by curative treatment by surgery with or without chemotherapy (induction or adjuvant) or by chemoradiotherapy
* Inoperable patients treated by exclusive radiotherapy
* A whole-body (skull base to mid thighs) FDG-PET or a combined FDG-PET/CT on a dedicated machine, performed before any anticancer treatment
* FDG-PET or combined FDG-PET/CT has to be previously standardised according to the procedure described in appendix IV
* Written informed consent
* Accessibility to follow-up
* Age > 18 years

Exclusion Criteria:

* Prior anticancer treatment (surgery, radiotherapy or chemotherapy)
* Stage IV NSCLC
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix and cured malignant tumour (more than 5-year disease free interval)
* Uncontrolled diabetes mellitus (fast glycaemia above 130 mg/dl)
* Pregnancy and lactating woman
* Unavailability to send a copy of the PET or PET-CT (DICOM format) to the data centre

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with non metastatic non small cell lung carcinoma, treated in the participating centres with curative intent
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2008-07; Primary Completion 2021-01 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Survival | Survival will be dated from the date of PET scan

SECONDARY OUTCOMES:
Progression-free survival | Period between the date of PET scan and the date of first progression or death

OTHER OUTCOMES:
discriminant value of 18F-FDG uptake for survival and for PFS | dated from PET examination

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, Study Chair — European Lung Cancer Working Party
Locations (6):
- Belgium (6):
  - Department of Pneumology RHMS Hôpital de la Madeleine, Ath
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Department of Pneumology CHU Charleroi, Charleroi
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - Department of Pneumology Centre Hospitalier de Mouscron, Mouscron

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Click here for more information on the protocol — http://www.elcwp.org